CLINICAL TRIAL: NCT05089318
Title: Curcuminoids and Boswellia Serrata Extracts Combination Decreases Hand Joint Discomfort : Results From a Belgian Real-Life Experience
Brief Title: Evaluation of Flexofytol® PLUS in Hand Joint Chronic Dyscomfort.
Status: Completed | Type: Observational
Sponsor: Tilman S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: FLEXOPAM
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-11

CONDITIONS: Hand Joint Discomfort
Keywords: Hand joint pain; curcumin; boswellia serrata; support to standard treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Flexofytol PLUS — 2 tablets in the morning and in the evening for minimum 6 weeks.

SUMMARY:
The purpose of this study is to evaluate the effect of curcuminoids and Boswellia serrata extracts combination (Flexofytol PLUS) in support to standard treatments during a 12-weeks period on hand pain on people with chronic hand joint discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Older dan 45 years old,
* With hand joint chronic discomfort,
* Regularly uses of paracetamol or NSAIDs to manage pain,
* Painful symptoms must have been present for more than 6 months,
* The patient assesses their pain on a visual pain scale and must be greater than 4 out of 10 over the last 48 hours.

Exclusion Criteria:

* Related to previous and associated treatments:

  * Corticosteroids injection in the 3 previous months, whatever the joint concerned,
  * Use of Slow-acting drugs for OA and/or dietary supplements taken within less than 6 months prior to the study (ex: chondroitin sulfate, diacerein, soy and avocado unsaponifiables, oxaceprol, granions de cuivre, glucosamine, phytotherapy or homeopathy for hand joint discomfort..),
  * Anticoagulant (coumarinic) treatment and heparin,
  * General corticotherapy in the 3 previous months,
  * Contraindication to paracetamol, curcumin, boswellia and NSAID's.
* Related to associated pathologies:

  * Patient suffering from serious associated illness (liver failure, kidney failure, non-controlled cardiovascular diseases...),
  * The patient has rheumatoid arthritis or gout,
  * The patient has a bile obstruction.
* Related to patient:

  * Pregnant or breastfeeding women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults above 45 years with chronic hand joint discomfort
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Pain using a Numerical Rating Scale (NRS) | 84 days
  Change from baseline of the mean pain over the last 48 hours evaluated by the patient on a 0 to 10 scale ( 0= no pain and 10=maximal pain)

CONTACTS AND LOCATIONS:
Overall Officials: Yvan Dierckxsens, Study Director — Tilman S.A.
Locations (2):
- Belgium (2):
  - Yves Henrotin, Boncelles, Liège
  - Yves Henrotin, Boncelles